CLINICAL TRIAL: NCT01943890
Title: Establishment and Implementation of Nebulised High Volumes of Hypertonic Saline in Cystic Fibrosis Patients
Brief Title: High Volumes of Hypertonic Saline and Chest Physiotherapy in CF Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009/2125
Record Dates: First submitted 2012-05-16; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Cystic Fibrosis
Keywords: Hypertonic saline; Lung physiotherapy
MeSH Terms: conditions — Cystic Fibrosis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physiotherapy and hypertonic saline (Experimental): Chest physiotherapy integrated with inhalation of hypertonic saline
  Interventions: Device: Hypertonic saline; Procedure: Physiotherapy

INTERVENTIONS:
Device: Hypertonic saline — 1 mmol/ml hypertonic saline given from (small children) 1,5 ml in 3 positions twice daily increasing to (children) 2 ml in 3 positions twice daily and up to (adults) 3 ml in 3 positions twice daily
Procedure: Physiotherapy

SUMMARY:
Background Nebulised hypertonic saline (HS) is an established basic airway clearance treatment in Cystic Fibrosis (CF). However, there is scarce evidence regarding the practical implementation and administration of different HS volumes, including physiotherapy and aspects of breathing pattern.

The aim of the study was to implement standardised and age-adjusted nebulised volumes of hypertonic saline in cystic fibrosis patients, included in physiotherapy and lung drainage techniques.

DETAILED DESCRIPTION:
Aims: To establish a safe, efficient routine for implementation of HS in daily treatment and to investigate the efficiency and tolerance of high volumes of HS integrated with chest physiotherapy.

HS was given twice daily with volumes of 4,5 ml in children aged 0-5 years, 6 ml at age 6-16 years and 9 ml at age > 16 years. The protocol included guidance of standardized breathing pattern, upright and sideways positioning and voluntary cough.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis

Exclusion Criteria:

* Non-adherence

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Tolerance and safety of high volumes of inhaled hypertonic saline measured by forced expiratory volume at one second | 24 months

SECONDARY OUTCOMES:
Implementation of nebulised high volumes of hypertonic saline in cystic fibrosis patients | 24 months
  Establishment of a standardized routine of nebulised high volumes of hypertonic saline including chest physiotherapy in cystic fibrosis patients

CONTACTS AND LOCATIONS:
Overall Officials: Stian Hammer, Principal Investigator — Dept. of Physiotherapy, Haukeland University Hospital, Bergen, Norway
Locations (1):
- Dept. of Thoracic Medicine, Haukeland University Hospital, Bergen, Norway